CLINICAL TRIAL: NCT00467233
Title: A Randomized, Rater-blinded, Split-face Comparison of the Efficacy of 30 % Salicylic Acid Peel vs. Q-switched Nd:Yag Laser for the Treatment of Melasma.
Brief Title: Study of Acid Peel and Laser for the Treatment of Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU679
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Laser Treatment
  Interventions: Procedure: Laser Treatment
- 2 (Experimental): Acid peel
  Interventions: Procedure: Acid Peel

INTERVENTIONS:
Procedure: Laser Treatment — Laser treatment to half of the face at each study visit
  Arms: 1
Procedure: Acid Peel — Acid peel to half of the face at each study visit
  Arms: 2

SUMMARY:
The objective of this study is to evaluate laser treatment and acid peel for the treatment of melasma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of laser treatment and acid peel for the treatment of melasma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melasma lesion measuring at least 4 square centimeters.
* Age 18-75 years.
* Good health.
* Willingness and ability to understand and provide informed consent for participation in the study.
* Ability to communicate with the investigator.
* Must be willing to forgo other treatment options for melasma during the course of the study.

Exclusion Criteria:

* Inability to understand the protocol or to give informed consent.
* Mental illness.
* Under 18 years of age and over 75 years of age.
* Laser treatment in the last 6 months before enrollment.
* Isotretinoin within the past year.
* Lidocaine allergy.
* History of herpes simplex viral infection.
* Concurrent active disease to facial area (i.e acne).
* Bleeding disorder.
* History of abnormal wound healing.
* History of abnormal scarring.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
MASI | 20 weeks

SECONDARY OUTCOMES:
Safety | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States